CLINICAL TRIAL: NCT04343209
Title: Ammonia N-13 Myocardial Blood Flow Absolute Quantification by Positron Emission Tomography in Patients With Known or Suspected Coronary Artery Disease (Ammonia MAP)
Brief Title: Ammonia N-13 Myocardial Blood Flow Absolute Quantification by PET in Patients With Known or Suspected CAD (Ammonia MAP)
Status: Completed | Type: Observational
Sponsor: Ionetix Corporation (Industry)
Responsible Party: Sponsor
Other Study IDs: Pro00042364
Record Dates: First submitted 2020-04-07; First posted 2020-04-13 (Actual); Last update posted 2024-09-05 (Actual); Status verified 2024-09

CONDITIONS: Myocardial Ischemia; Coronary Disease; Coronary Artery Disease; Heart Diseases; Cardiovascular Diseases; Arteriosclerosis; Arterial Occlusive Diseases; Vascular Diseases
Keywords: Ammonia N-13; Positron Emission Tomography; Myocardial Blood Flow; MBF; Myocardial Perfusion; Ammonia N 13 Injection, USP; Coronary Artery Disease
MeSH Terms: conditions — Myocardial Ischemia; Coronary Disease; Coronary Artery Disease; Heart Diseases; Cardiovascular Diseases; Arteriosclerosis; Arterial Occlusive Diseases; Vascular Diseases | interventions — Injections, Intravenous

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Individuals with confirmed or suspected cardiovascular disease: Individuals in this group will undergo myocardial perfusion imaging, utilizing Ammonia N-13 PET imaging agent. Each individual will receive two intravenous injections of Ammonia N-13 in accordance with site imaging protocol.
  Interventions: Diagnostic Test: Myocardial Perfusion Imaging Study; Drug: AMMONIA N-13 37.5 mCi in 1 mL INTRAVENOUS INJECTION [Ammonia N 13]

INTERVENTIONS:
Diagnostic Test: Myocardial Perfusion Imaging Study — Evaluation of myocardial perfusion via PET imaging agent
Drug: AMMONIA N-13 37.5 mCi in 1 mL INTRAVENOUS INJECTION [Ammonia N 13] — Cardiac PET imaging agent

SUMMARY:
This study is being conducted to provide access to and collect test data for an established nuclear medicine diagnostic imaging test called Positron Emission Tomography (PET), using a specific radioactive drug called Ammonia N-13 (Ammonia), referred to simply as an Ammonia PET scan, which is used to visualize the blood flow through the blood vessels and into the heart muscle in order to identify areas of restricted blood flow within the heart. The scanner used in this study may be a stand-alone PET scanner or a PET/CT scanner, which combines the PET scanner and a Computed Tomography (CT) scanner into a single device. Unless otherwise stated in this consent form, the term PET will be used to refer to both stand-alone PET and PET/CT scanners. While physicians have used the Ammonia PET test for many years to visualize (image) the blood flow into the heart muscle (perfusion), it is now possible to also measure the flow of blood into the heart muscle. Research studies have demonstrated clinical value in reviewing the measured blood flow values in addition to reviewing the perfusion images of blood flow into the heart muscle. Therefore, this study will establish a database of a large number of Ammonia PET measured blood flow values to serve as a future reference.

DETAILED DESCRIPTION:
This is a prospective, multicenter database that will be populated by sites utilizing N-13 Ammonia and sponsored by Ionetix. Each site with access to N-13 produced under an investigational new drug (IND) application will be eligible to participate. Once the site is activated, the site will enroll patients into the database that are scheduled for clinically indicated PET-MPI with N-13 (as determined by their treating physicians). PET-MPI perfusion, MBF, percent ischemia, pharmacologic stress agent, and gated left ventricular ejection fraction/function values will be collected when available, in an anonymous fashion and uploaded into the database. All patient health identifiers (PHI) will be removed prior to upload. No procedures additional to those clinically indicated will be performed for the purposes of this study.

ELIGIBILITY:
Inclusion Criteria:

Adults ≥18 able to give informed consent.

Clinical indication for PET-MPI as determined by the subject's treating physician

Exclusion Criteria:

Any clinical contraindication for pharmacologic stress testing per ASNC/SNMMI/ACC myocardial perfusion imaging guidelines when stress perfusion imaging is required clinically.

Inability or unwilling to give informed consent

Pregnant subjects

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Individuals with confirmed or suspected cardiovascular disease
Sampling Method: Non-Probability Sample
Enrollment: 170 (Actual)
Dates: Start 2020-09-14 (Actual); Primary Completion 2024-08-16 (Actual); Study Completion 2024-08-16 (Actual)

PRIMARY OUTCOMES:
Establish the N-13 measured MBF (ml/g/min) value range | an estimated average of 2 hours
  Non-invasive measurements of myocardial blood flow (MBF) in milliliter/minute/gram using PET/CT or PET scanner will be compared to invasive cardiac angiography values (current gold standard). MBF values are obtained using image-derived time activity curves from the left ventricular blood and myocardial tissue regions. These values represent radiotracer exchange between the blood and the tissue over time. The rate of radiotracer uptake into the myocardial tissue provides an estimate of MBF. Processing software will then use the time-activity curves to calculate MBF at rest and at stress.

CONTACTS AND LOCATIONS:
Overall Officials: Joseph Oliverio, Study Director — Ionetix Corporation
Locations (5):
- United States (5):
  - Doral Imaging Institute, LLC dba CIRA, Miami, Florida
  - Doral Imaging Institute, LLC DBA CIRA Miami Beach, Miami Beach, Florida
  - Adler Institute for Advanced Imaging, Jenkintown, Pennsylvania
  - UPMC, Pittsburgh, Pennsylvania
  - Molecular Imaging Technologies, El Paso, Texas

REFERENCES:
- [Result] Araujo LI, Lammertsma AA, Rhodes CG, McFalls EO, Iida H, Rechavia E, Galassi A, De Silva R, Jones T, Maseri A. Noninvasive quantification of regional myocardial blood flow in coronary artery disease with oxygen-15-labeled carbon dioxide inhalation and positron emission tomography. Circulation. 1991 Mar;83(3):875-85. doi: 10.1161/01.cir.83.3.875. PMID 1900224
- [Result] Bergmann SR, Herrero P, Markham J, Weinheimer CJ, Walsh MN. Noninvasive quantitation of myocardial blood flow in human subjects with oxygen-15-labeled water and positron emission tomography. J Am Coll Cardiol. 1989 Sep;14(3):639-52. doi: 10.1016/0735-1097(89)90105-8. PMID 2788669
- [Result] Sdringola S, Johnson NP, Kirkeeide RL, Cid E, Gould KL. Impact of unexpected factors on quantitative myocardial perfusion and coronary flow reserve in young, asymptomatic volunteers. JACC Cardiovasc Imaging. 2011 Apr;4(4):402-12. doi: 10.1016/j.jcmg.2011.02.008. PMID 21492816
- [Result] Merlet P, Mazoyer B, Hittinger L, Valette H, Saal JP, Bendriem B, Crozatier B, Castaigne A, Syrota A, Rande JL. Assessment of coronary reserve in man: comparison between positron emission tomography with oxygen-15-labeled water and intracoronary Doppler technique. J Nucl Med. 1993 Nov;34(11):1899-904. PMID 8229231
- [Result] Kern MJ, Bach RG, Mechem CJ, Caracciolo EA, Aguirre FV, Miller LW, Donohue TJ. Variations in normal coronary vasodilatory reserve stratified by artery, gender, heart transplantation and coronary artery disease. J Am Coll Cardiol. 1996 Nov 1;28(5):1154-60. doi: 10.1016/S0735-1097(96)00327-0. PMID 8890809
- [Result] Gewirtz H, Fischman AJ, Abraham S, Gilson M, Strauss HW, Alpert NM. Positron emission tomographic measurements of absolute regional myocardial blood flow permits identification of nonviable myocardium in patients with chronic myocardial infarction. J Am Coll Cardiol. 1994 Mar 15;23(4):851-9. doi: 10.1016/0735-1097(94)90629-7. PMID 8106689
- [Result] Rivas F, Cobb FR, Bache RJ, Greenfield JC Jr. Relationship between blood flow to ischemic regions and extent of myocardial infarction. Serial measurement of blood flow to ischemic regions in dogs. Circ Res. 1976 May;38(5):439-47. doi: 10.1161/01.res.38.5.439. PMID 1269083
- [Result] Renaud JM, Yip K, Guimond J, Trottier M, Pibarot P, Turcotte E, Maguire C, Lalonde L, Gulenchyn K, Farncombe T, Wisenberg G, Moody J, Lee B, Port SC, Turkington TG, Beanlands RS, deKemp RA. Characterization of 3-Dimensional PET Systems for Accurate Quantification of Myocardial Blood Flow. J Nucl Med. 2017 Jan;58(1):103-109. doi: 10.2967/jnumed.116.174565. Epub 2016 Aug 18. PMID 27539843
- [Result] Murthy VL, Naya M, Foster CR, Hainer J, Gaber M, Di Carli G, Blankstein R, Dorbala S, Sitek A, Pencina MJ, Di Carli MF. Improved cardiac risk assessment with noninvasive measures of coronary flow reserve. Circulation. 2011 Nov 15;124(20):2215-24. doi: 10.1161/CIRCULATIONAHA.111.050427. Epub 2011 Oct 17. PMID 22007073
- [Result] Ziadi MC, Dekemp RA, Williams KA, Guo A, Chow BJ, Renaud JM, Ruddy TD, Sarveswaran N, Tee RE, Beanlands RS. Impaired myocardial flow reserve on rubidium-82 positron emission tomography imaging predicts adverse outcomes in patients assessed for myocardial ischemia. J Am Coll Cardiol. 2011 Aug 9;58(7):740-8. doi: 10.1016/j.jacc.2011.01.065. PMID 21816311